CLINICAL TRIAL: NCT05003206
Title: Multimodal Magnetic Resonance Imaging Studying the Mechanism and Predicting the Outcome After Deep Brain Stimulation in Patients With Parkinson's Disease
Brief Title: Predictive Value of Multimodal MRI in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Director of Department of Radiology, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Multimodal MRI DBS-PD
Record Dates: First submitted 2021-07-01; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Parkinson's Disease; Magnetic Resonance Imaging; Deep Brain Stimulation
Keywords: Subthalamic nucleus deep brain stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD,DBS (Experimental): Patients with idiopathic PD before and after DBS surgery
  Interventions: Other: Functional magnetic resonance imaging; Device: Deep Brain Stimulation

INTERVENTIONS:
Other: Functional magnetic resonance imaging — Preoperative and postoperative functional magnetic resonance imaging (fMRI) scanning. fMRI is a new neuroimaging method. Its principle is to use magnetic resonance imaging to measure the changes of hemodynamics caused by neuronal activity.
Device: Deep Brain Stimulation — For PD patients treated with DBS, the neurologist will turn off the stimulator before MRI scan

SUMMARY:
Deep brain stimulation (DBS) is recognized as the most safe and effective neurosurgical method for the treatment of advanced Parkinson's disease. However, the mechanism of relieving motor and non-motor symptoms of Parkinson's disease has not been fully clarified, and the prognosis is significantly different. This study is based on multimodal MRI technique to clarify the mechanism of DBS in relieving motor and non-motor symptoms of Parkinson's disease, and to explore imaging indicators that can predict prognosis, so as to guide the individual and accurate treatment of Parkinson's disease (PD).

DETAILED DESCRIPTION:
1. Preoperative and postoperative multimodal MRI scanning 1) equipment: 3TGE 750 MRI 2) sequence: resting state fMRI, DTI, 3DTI, ESWAN, ASL 3) scan status: drug shutdown period ( discontinuation of drugs for Parkinson's disease for at least 12 hours), for patients who can not adhere to MRI scanning after drug withdrawal. Record the dosage of drugs before scanning
2. Evaluation of motor and non-motor symptoms: pre-operation and 1-year post-operation 1) motor symptoms: pre-operation medication opening and closing period. Postoperative medication off/stimulation off (Med-OFF/DBS-OFF);Med-ON/DBS-OFF;Med-OFF/DBS-ON;Med-ON/DBS-ON

   1. overall evaluation of motor function: MDS-UPRDS, H&Y stage
   2. balance: Berg balance scale
   3. dyskinesia: abnormal involuntary movement scale(AIMS)
   4. end-of-dose phenomenon: WOQ19 end-of-dose phenomenon questionnaire
   5. daily activity ability: SCHWAB&ENGLAND daily activity scale 2) non-motor symptoms: preoperative drug shutdown period. Postoperative drug shutdown / DBS opening

   <!-- -->

   1. Cognitive function: Mini Mental State Examination scale (MMSE), Montreal Cognitive Assessment scale (MoCA)
   2. emotion: Hamilton Depression scale (HAMD), Hamilton anxiety scale (HAMA)
   3. Sleep: PD Sleep scale (PDSS), Appleworth sleepiness scale (ESS), REM Sleep Behavioral Disorder questionnaire-Hong Kong (RBDQ-HK)
   4. pain: King Parkinson's disease pain scale (KPPS)
   5. fatigue: fatigue severity scale (FSS)
   6. autonomic nervous function assessment: autonomic nervous scale (SCOPA-AUT) h) quality of life: 39 items Parkinson's disease quality of life questionnaire (PDQ-39) 3.other records: changes in type, dose and mode of use of drugs. Daily equivalent dose of levodopa (tomlinson2010 conversion)

ELIGIBILITY:
Inclusion Criteria:

* Patient with Parkinson's disease
* age< 70 years
* Underwent bilateral STN-DBS or not
* Having complete medical history and clinical follow up
* All MRI examination performed according to study protocol
* Imaging data can be processed
* Signed informed consent obtained from the patient or patient's legally authorized representative;

Exclusion Criteria:

* Parkinson-plus syndrome or secondary parkinsonism
* Patients with severe mental disorders such as psychosis, liver and kidney dysfunction, poor blood pressure or blood glucose control, severe depression and substance abuse, low IQ, and acute phase of severe stroke with definite limb dysfunction should also be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-19 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics of patients | 1 to 2 years
  Age at onset; age at surgery; disease duration; level of education; comorbidities (e.g. hypertension and diabetes mellitus); parkinsonism subtype; period of motor fluctuations; time from motor fluctuations to surgery; cigarette smoking
Percentage of improvement in motor aspects (after 12 months of stimulation) | 1 to 3 years
  (UPDRS III 12 months - UPDRS III baseline)/UPDRS III baseline where UPDRS III 12 months means the score of this test in "medication off , stimulation on" condition at 12 months after implant, while UPDRS III baseline means the score of this test in "medication off " condition.The clinical outcome, or degree of symptom benefit, was defined as a ≥50% improvement on a disease severity rating scale

SECONDARY OUTCOMES:
other records: | 1 to 3 years
  Changes in type, dose and mode of use of drugs. Daily equivalent dose of levodopa (tomlinson2010 conversion)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No